CLINICAL TRIAL: NCT03892538
Title: Correlation Between Blood Pressure, Heart Rate and Plasma Corticotropin, Cortisol Under Surgical Skin Incision
Status: Completed | Type: Observational
Sponsor: JingCang (Other)
Responsible Party: Sponsor-Investigator, JingCang, Director, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Other Study IDs: B2018-288R
Record Dates: First submitted 2019-03-13; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2018-10

CONDITIONS: Stress, Psychological
Keywords: Stress; Blood pressure; Heart rate; Corticotropin; Cortisol
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective observational study was conducted to analyze the correlation between systolic blood pressure, diastolic blood pressure, mean arterial pressure，heart rate and plasma corticotropin, cortisol during surgical skin incision.

DETAILED DESCRIPTION:
The elements of general anesthesia include sedation, analgesia and muscle relaxation, while the essence of intraoperative pain in patients under general anesthesia is the body's unconscious response to tissue damage, namely the stress response.Stress response is a series of hormonal and metabolic changes produced by the body in response to nociceptive stimuli. It is part of the systemic response to injury and includes a wide range of endocrine, immunological and hemodynamic effects.Operation as well as the modern medicine common disease treatment, as a harmful stimulation, can cause the body strong stress reaction, reaction and duration and the size of the surgery is often proportional to the damage degree, its mechanism mainly include the activation of the sympathetic nervous system, adrenocorticotropic hormone (ACTH), growth hormone, vasopressin (AVP), cortisol and aldosterone and a series of hypothalamus pituitary adrenal axis hormone changes, insulin resistance and stress hyperglycemia, IL - 1, IL - 6, TNF alpha, such as the change of cytokines,And the increase in acute phase reactions such as acute response phase protein (CRP).As a protective response, stress response can mobilize the energy stored in the body when the body is injured, and help the body survive in harsh environment.But now a good perioperative management environment means that patients can be adequately nourished even after surgery.In this case, excessive stress response leads to preoperative anxiety of patients, the occurrence of adverse events in the intraoperative central blood vessels, and the occurrence of postoperative complications.In surgical patients, many systems, including the brain, are negatively affected by stress hormones.Perioperative acute stress can lead to post-traumatic stress disorder, depression, postoperative fatigue, chronic pain, and cognitive decline in elderly patients.Perioperative hyperglycemia and insulin resistance are closely related to postoperative infection and cardiovascular events, and may prolong hospital stay.Perioperative stress response will also damage the immune function of patients, which is mainly manifested as inhibition of natural killer cell function and inhibition of innate immune function response, which brings concerns about postoperative infection and tumor recurrence of patients.Anesthesia can inhibit the intraoperative stress of patients to a certain extent. Different anesthesia drugs and anesthesia methods can be selected for the same operation.Dexmedetomidine has dose-dependent sedative, analgesic, anti-anxiety and hypnotic effects. It can reduce serum s-100 protein, lipid peroxidation product malondialdehyde (MDA), raise the level of hyper oxide dismutase (SOD), and reduce TNF-, il-1, il-6 and other pro-inflammatory mediators.Fentanyl, rui fentanyl, sufentanil opioids can inhibit the hypothalamus pituitary adrenal axis, decrease the plasma levels of stress hormones, but this does not mean that the investigators can in the art of unlimited increase the drug, also want to consider the stability of hemodynamics, respiratory depression caused by delayed awakening, postoperative nausea and vomiting, postoperative itching and postoperative recovery of gastrointestinal, etc.;Epidural anesthesia with segmental sympathetic nerve blocking effect, in the chest surgery, general anesthesia compound epidural block than all by intravenous anesthesia, the patient's heart rate, blood pressure, mean arterial pressure, such as index significantly more smoothly, catecholamine levels in peripheral blood, the incidence of postoperative adverse events also significantly reduced.Real-time monitoring of the intraoperative stress level of patients is helpful for the anesthesiologist to determine the depth of anesthesia and guide the intraoperative anesthesia medication.There are many ways to monitor the level of intraoperative stress in patients.Surgical volume index (SPI) is used to monitor the pain-analgesic balance during general anesthesia through heartbeat interval and pulse wave amplitude measured by light.Skin pain conductance meter (SCA) assesses the size and pain of nociceptive stimulation through sweating and skin conductance.The pupil pain index (PPI) monitors intraoperative pain by measuring changes in pupil size caused by nociceptive stimulation.All of these indicators were used to monitor the intraoperative stress level through sympathetic or parasympathetic nerve activity. However, the intraoperative acute stress response was related to the state of high adrenocorticotropin and high cortisol. Currently, there is no index to evaluate the intraoperative pain of patients based on the change of intraoperative stress hormone level.However, the changes of stress hormones must be detected by laboratory tests. Therefore, whether the changes of stress hormones can be estimated by the blood pressure and heart rate that the investigators routinely monitor during the operation, so as to provide a research direction for us to establish the intraoperative pain monitoring method with stress hormones as the evaluation standard.In summary, this clinical study analyzed the relationship between the changes of systolic blood pressure, diastolic blood pressure, mean arterial pressure and heart rate under surgical curettage stimulation and the changes of plasma adrenocorticotrophin and cortisol through prospective observational studies, and found out the indexes that could reflect the changes of stress hormones during the operation.

ELIGIBILITY:
Inclusion Criteria:

* the ASA score was from grade I to III,
* aged 18-80 years

Exclusion Criteria:

* adrenal gland related diseases
* immune system related diseases
* severe cardiovascular and cerebrovascular diseases,
* severe liver and kidney dysfunction
* refuse to participate in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The enrolled patients were mainly male and the type of surgery was open upper abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | Change from skin incision till 10 minutes after skin incision
  mmHg
diastolic blood pressure | Change from skin incision till 10 minutes after skin incision
  mmHg
mean arterial pressure | Change from skin incision till 10 minutes after skin incision
  mmHg
heart rate | Change from skin incision till 10 minutes after skin incision
  bpm
corticotropin | Change from skin incision till 10 minutes after skin incision
  plasma concentration，pg/ml
cortisol | Change from skin incision till 10 minutes after skin incision
  plasma concentration，nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Jing Cang, PHD, Study Director — Director
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data not yet collated

REFERENCES:
- [Background] Huiku M, Uutela K, van Gils M, Korhonen I, Kymalainen M, Merilainen P, Paloheimo M, Rantanen M, Takala P, Viertio-Oja H, Yli-Hankala A. Assessment of surgical stress during general anaesthesia. Br J Anaesth. 2007 Apr;98(4):447-55. doi: 10.1093/bja/aem004. Epub 2007 Feb 28. PMID 17329347
- [Background] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999
- [Background] Pan YS, Hu YF, Tian FB, Xu K. Effects of epidural preemptive analgesia on stress reaction in retroperitoneal laparoscopic adrenalectomy surgery: a randomized controlled study. Int J Clin Exp Med. 2015 Jun 15;8(6):9862-8. eCollection 2015. PMID 26309669
- [Background] McEwen BS. The neurobiology of stress: from serendipity to clinical relevance. Brain Res. 2000 Dec 15;886(1-2):172-189. doi: 10.1016/s0006-8993(00)02950-4. PMID 11119695
- [Background] Rodrigues SM, LeDoux JE, Sapolsky RM. The influence of stress hormones on fear circuitry. Annu Rev Neurosci. 2009;32:289-313. doi: 10.1146/annurev.neuro.051508.135620. PMID 19400714
- [Background] Borsook D, George E, Kussman B, Becerra L. Anesthesia and perioperative stress: consequences on neural networks and postoperative behaviors. Prog Neurobiol. 2010 Dec;92(4):601-12. doi: 10.1016/j.pneurobio.2010.08.006. Epub 2010 Aug 19. PMID 20727935
- [Background] Sato H, Carvalho G, Sato T, Lattermann R, Matsukawa T, Schricker T. The association of preoperative glycemic control, intraoperative insulin sensitivity, and outcomes after cardiac surgery. J Clin Endocrinol Metab. 2010 Sep;95(9):4338-44. doi: 10.1210/jc.2010-0135. Epub 2010 Jul 14. PMID 20631016
- [Background] Ljungqvist O. Jonathan E. Rhoads lecture 2011: Insulin resistance and enhanced recovery after surgery. JPEN J Parenter Enteral Nutr. 2012 Jul;36(4):389-98. doi: 10.1177/0148607112445580. Epub 2012 May 10. PMID 22577121
- [Background] Nygren J. The metabolic effects of fasting and surgery. Best Pract Res Clin Anaesthesiol. 2006 Sep;20(3):429-38. doi: 10.1016/j.bpa.2006.02.004. PMID 17080694
- [Background] Liu Z, Jiang M, Zhao J, Ju H. Circulating tumor cells in perioperative esophageal cancer patients: quantitative assay system and potential clinical utility. Clin Cancer Res. 2007 May 15;13(10):2992-7. doi: 10.1158/1078-0432.CCR-06-2072. PMID 17505001
- [Background] Li Y, Liu S. The Effect of Dexmedetomidine on Oxidative Stress Response Following Cerebral Ischemia-Reperfusion in Rats and the Expression of Intracellular Adhesion Molecule-1 (ICAM-1) and S100B. Med Sci Monit. 2017 Feb 17;23:867-873. doi: 10.12659/msm.899855. PMID 28212354
- [Background] Anand KJ, Sippell WG, Aynsley-Green A. Randomised trial of fentanyl anaesthesia in preterm babies undergoing surgery: effects on the stress response. Lancet. 1987 Jan 31;1(8527):243-8. doi: 10.1016/s0140-6736(87)90065-1. PMID 20928962
- [Background] Anand KJ, Hickey PR. Halothane-morphine compared with high-dose sufentanil for anesthesia and postoperative analgesia in neonatal cardiac surgery. N Engl J Med. 1992 Jan 2;326(1):1-9. doi: 10.1056/NEJM199201023260101. PMID 1530752
- [Background] Li C, Xu M, Wu Y, Li YS, Huang WQ, Liu KX. Limb remote ischemic preconditioning attenuates lung injury after pulmonary resection under propofol-remifentanil anesthesia: a randomized controlled study. Anesthesiology. 2014 Aug;121(2):249-59. doi: 10.1097/ALN.0000000000000266. PMID 24743579
- [Background] Hopf HB, Weissbach B, Peters J. High thoracic segmental epidural anesthesia diminishes sympathetic outflow to the legs, despite restriction of sensory blockade to the upper thorax. Anesthesiology. 1990 Nov;73(5):882-9. doi: 10.1097/00000542-199011000-00015. PMID 2240678
- [Background] Freise H, Van Aken HK. Risks and benefits of thoracic epidural anaesthesia. Br J Anaesth. 2011 Dec;107(6):859-68. doi: 10.1093/bja/aer339. Epub 2011 Nov 4. PMID 22058144
- [Background] Sidiropoulou I, Tsaousi GG, Pourzitaki C, Logotheti H, Tsantilas D, Vasilakos DG. Impact of anesthetic technique on the stress response elicited by laparoscopic cholecystectomy: a randomized trial. J Anesth. 2016 Jun;30(3):522-5. doi: 10.1007/s00540-016-2148-7. Epub 2016 Feb 16. PMID 26882921
- [Background] Ryu KH, Kim JA, Ko DC, Lee SH, Choi WJ. Desflurane reduces intraoperative remifentanil requirements more than sevoflurane: comparison using surgical pleth index-guided analgesia. Br J Anaesth. 2018 Nov;121(5):1115-1122. doi: 10.1016/j.bja.2018.05.064. Epub 2018 Jul 4. PMID 30336856
- [Background] Storm H. Changes in skin conductance as a tool to monitor nociceptive stimulation and pain. Curr Opin Anaesthesiol. 2008 Dec;21(6):796-804. doi: 10.1097/ACO.0b013e3283183fe4. PMID 18997532
- [Background] Sabourdin N, Diarra C, Wolk R, Piat V, Louvet N, Constant I. Pupillary Pain Index Changes After a Standardized Bolus of Alfentanil Under Sevoflurane Anesthesia: First Evaluation of a New Pupillometric Index to Assess the Level of Analgesia During General Anesthesia. Anesth Analg. 2019 Mar;128(3):467-474. doi: 10.1213/ANE.0000000000003681. PMID 30198934